CLINICAL TRIAL: NCT03741010
Title: Belviq Tablet® Post Marketing Surveillance Protocol
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: IlDong Pharmaceutical Co Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: ID-BVQ-401
Record Dates: First submitted 2018-11-12; First posted 2018-11-14 (Actual); Last update posted 2018-11-26 (Actual); Status verified 2018-08

CONDITIONS: Weight Loss
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Post-marketing surveillance of Lorcaserin

DETAILED DESCRIPTION:
Lorcaserin(Belviq) is a selective 5-hydroxytryptamine receptor agonist, witch is used long term for weight loss in those who are obese. Lorcaserin was approved in 2015 the Republic of Korea for weigh loss in those who are obese. A post-marketing surveillance was conducted following the approval to obtain data on the safety and efficacy of lorcaserin for weigh loss in real-world practice.

ELIGIBILITY:
Inclusion Criteria:

Subjects who use the drug as an adjuvant therapy of diet therapy and kinesitherapy for weight control are selected.

1. Obese patients whose body mass index (BMI) is ≧30 kg/m2.
2. Overweight patients whose body mass index(BMI) is ≧27 kg/m2 and who have other risk factors(e.g. hypertension, dyslipidemia, type II diabetes mellitus)

Exclusion Criteria:

1. Patients with a hypersensitivity reaction to the drug or the ingredient of the drug
2. Female patients of childbearing potential and pregnant or lactating women
3. Patients taking another weight control drug
4. Patients with the medical history of drug abuse

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: residents of Korea, in real-world practice
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2015-02-02 (Actual); Primary Completion 2021-02-01 (Estimated); Study Completion 2021-02-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse event after this drug administration in general medical | 12 weeks
  Any adverse events occurred after this drug dosing will be recorded. Description of adverse event(s) including type of adverse event(s), onset/end date, severity, action taken, causal relationship to the drug and investigator's view on the adverse event(s) will be captured, whether it is related to the drug or not and until follow up visit more than 1 time during the surveillance period.
  Lab abnormalities and changes in vital signs are considered to be adverse events only if they result in discontinuation from the study, necessitate therapeutic medical intervention, and/or if the investigator considers them to be adverse events.

SECONDARY OUTCOMES:
The change from baseline to week 12 in the Body Mass Index(BMI) | 12 weeks
  BMI is measured before administration of the drug and within 12 weeks after administration.

IPD SHARING:
Plan to Share IPD: Undecided